CLINICAL TRIAL: NCT01963130
Title: Does Vildagliptin Affect Portal Vein Pressure In Patients With Type 2 Diabetes Mellitus? A Cross Sectional Study
Status: Completed | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Cumali Karatoprak, MD, Bezmialem Vakif University
Other Study IDs: ISRCTN73824458
Record Dates: First submitted 2013-10-10; First posted 2013-10-16 (Estimated); Last update posted 2013-10-16 (Estimated); Status verified 2013-10

CONDITIONS: Drug Mechanism; Drug Usage
Keywords: Vildagliptin; Portal Vein Pressure; Hepatosteatosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- drug (metformin and gliclazide): The first group (Group 1) consisted of patients that used metformin (1000 mg bid) and gliclazide (60 mg qd).
- drug (metformin, gliclazide and vildagliptin): The second group (Group 2) consisted of patients that used vildagliptin (50 mg bid) in addition to the same amount of metformin and gliclazide since their HbA1c were detected 7 % or over.

SUMMARY:
This study investigated how vildagliptin (a di-peptidyl peptidase 4 inhibitor) affects portal vein pressure and hepatosteatosis in patients with type 2 diabetes mellitus.

DETAILED DESCRIPTION:
Group 1 used metformin (1000 mg bid) and gliclazide (60 mg qd); Group 2 used the same amounts of metformin and gliclazide, with the addition of vildagliptin (50 mg bid). The patients were prospectively assigned to each of these two groups for the purpose of this study. Using Doppler ultrasound, all cases were measured for portal vein flow velocity, portal vein flow and portal vein diameter. Degree of hepatosteatosis was also recorded.

ELIGIBILITY:
Inclusion Criteria:

-type 2 DM cases and at least 3 months used the same drugs (metformin and gliclazide or metformin and gliclazide and vildagliptin)

Exclusion Criteria:

* used alcohol and cigarettes
* chronic liver disease,
* chronic renal failure,
* active infection
* patients using certain drugs which may affect portal pressure such as propronalol,
* calcium channel blockers,
* angiotensin-converting enzyme inhibitors,
* angiotensin receptor blockers and isosorbit monohydrate

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: type 2 Diabetes Mellitus (DM)
Sampling Method: Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2012-07; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
This study investigated the effect of the used type 2 DM drug, vildagliptin, a DPP-4 inhibitor, on portal hemodynamics. | at least 3 month (mean 7.8 months)
  This study investigated how vildagliptin (a di-peptidyl peptidase 4 inhibitor) affects portal vein pressure in patients with type 2 diabetes mellitus. Portal vein flow velocity, portal vein flow, and portal vein diameter of all cases were measured by Doppler ultrasound in both groups.

SECONDARY OUTCOMES:
This study investigated the effect of the used type 2 DM drug, vildagliptin, a DPP-4 inhibitor, on hepatosteatosis. | followed for at least 3 months (mean 7.8 months)
  Patients were examined in the left decubitus position with a Logiq 9 Review (GE, Milwaukee, WI, USA) ultrasound device and a 3.5-mHz convex transducer probe was used. Gray scale and color Doppler features were used. All segments of the liver were examined and the presence and degree of hepatosteatosis was recorded

CONTACTS AND LOCATIONS:
Overall Officials: Cumali Karatoprak, MD, Study Director — Bezmialem VU
Locations (1):
- Bezmialem VU, Istanbul, Turkey (Türkiye)